CLINICAL TRIAL: NCT01154686
Title: Working Memory Training in College Students With ADHD/LD
Brief Title: Working Memory Training in College Students With Attention-Deficit Hyperactivity Disorder/Learning Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Rachel Gropper, OISE/University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23977
Record Dates: First submitted 2010-04-14; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cogmed — The Cogmed Working Memory Training Program will be used as the experimental program because of preliminary evidence indicating its effectiveness in enhancing WM and reducing behavioural symptoms of inattention/hyperactivity in children. This software-based training program was designed to improve WM abilities, particularly in children with ADHD or severe attention problems. Training is implemented with a software program (RoboMemo©). It includes a set of auditory verbal and visual-spatial WM tasks presented via computer. All tasks involve: maintenance of simultaneous mental representations of multiple stimuli, unique sequencing of stimulus order in each trial and progressive adaptation of difficulty level as a function of individual performance.

SUMMARY:
The overall objective of the current study is to determine whether computerized Working Memory (WM) training will enhance WM capacity in college students with Attention Deficit Hyperactivity Disorder (ADHD)/Learning Disabilities (LD). There are also three additional objectives. The first is to determine whether improvements in WM will generalize to secondary outcome tasks, such as inhibitory control and planning. The second objective is to examine whether WM training will also ameliorate ADHD symptoms of inattention and hyperactivity. The last objective is to investigate whether improvements will be maintained at a two month follow-up period.

It is expected that the computerized WM training program will enhance WM capacity in college students with ADHD. In addition, it is believed that these increases in WM capacity will also lead to improvements in other executive functions. It is also hypothesized that WM training will lead to a reduction in ADHD symptomology. Lastly, these improvements should be maintained at three month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD/Learning Disability
* registered as a university student (full or part time)
* registered at accessibilities services
* taking at least one course

Exclusion Criteria:

* On a leave

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Paced Auditory Serial Addition Test (auditory verbal working memory measure) | within 120 days

SECONDARY OUTCOMES:
Cognitive Failures Questionnaire | within 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gropper, MA, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada